CLINICAL TRIAL: NCT07282093
Title: An Open-Label, Phase 1 Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics of Olverembatinib
Brief Title: Pharmacokinetics of Olverembatinib in Participants With Hepatic Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Guangzhou Healthquest Pharma Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351XC107
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pharmacokinetic; Olverembatinib
Keywords: olverembatinib
MeSH Terms: interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: 6-8 participants with mild hepatic impairment. (Experimental)
  Interventions: Drug: Olverembatinib 20mg
- Group 2: 6-8 participants with normal hepatic function matched to Group 1 (Experimental)
  Interventions: Drug: Olverembatinib 20mg
- Group 3: 6-8 participants with moderate hepatic impairment (Experimental)
  Interventions: Drug: Olverembatinib 20mg
- Group 4: 6-8 participants with normal hepatic function matched to Group 3 (Experimental)
  Interventions: Drug: Olverembatinib 20mg
- Group 5: 6-8 participants with severe hepatic impairment (Experimental)
  Interventions: Drug: Olverembatinib 20mg
- Group 6: 6-8 participants with normal hepatic function matched to Group 5 (Experimental)
  Interventions: Drug: Olverembatinib 20mg

INTERVENTIONS:
Drug: Olverembatinib 20mg — orally after meal, single dose

SUMMARY:
This is a non-randomized, open-label, parallel, single-dose study to evaluate the pharmacokinetic profile of olverembatinib in participants with normal or impaired liver function.

DETAILED DESCRIPTION:
To evaluate the PK characteristics of olverembatinib in participants with mild hepatic impairment (Child-Pugh Class A), moderate hepatic impairment (Child-Pugh Class B), severe hepatic impairment (Child-Pugh Class C) and sex, age, and body weight-matched healthy participants with normal hepatic function, so as to provide a scientific basis for the appropriate dose and/or dosing interval adjustment in participants with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant voluntarily joins the study, signs the Informed Consent Form, and demonstrates good compliance.
2. Body Mass Index (BMI) between 18 and 30 kg/m² (inclusive), with male weight ≥ 50 kg and female weight ≥ 45 kg.
3. The investigator judges the participant suitable to participate in this study based on physical examination, vital signs, laboratory tests, and 12-lead electrocardiogram (ECG) examination.
4. Female participants of childbearing potential must agree to use effective contraception during the study and for 3 months after the study ends; must have a negative serum pregnancy test within 7 days prior to study enrollment; and must not be breastfeeding. Male participants must agree to use effective contraception during the study and for 3 months after the study ends.
5. Additional Criteria for Participants with hepatic impairment Only:

1. Chronic hepatic impairment due to viral hepatitis, alcoholic liver disease, autoimmune hepatitis, or other causes.

2. Hepatic impairment classified as Child-Pugh Class A, B, or C. 3. Coagulation function: INR ≤ 2.5 without intervention with procoagulant drugs (after a 2-week washout period). Hematology: Neutrophils ≥ 1.0 × 10⁹/L, Hemoglobin ≥ 70 g/L, Platelets ≥ 30 × 10⁹/L. Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 5 times the Upper Limit of Normal (ULN); Total Bilirubin ≤ 5 × ULN.

4. Stable treatment for hepatic impairment, complications, and other concomitant diseases prior to study drug administration, with no need for dosage adjustment. Treatment for hepatic impairment must have been stable for at least 4 weeks.

Exclusion Criteria:

1. Drug-induced liver injury.
2. Any of the following conditions: history of liver transplantation; presence of acute or worsening liver injury due to any cause; liver failure; concurrent Grade 3/4 hepatic encephalopathy; active hepatocellular carcinoma lesions; severe esophageal or gastric varices or history of rupture and bleeding; severe/late-stage ascites or pleural effusion requiring paracentesis/thoracentesis and albumin supplementation; hepatorenal syndrome; or any other condition deemed by the investigator as unsuitable for study participation.
3. History of cholestasis, biliary tract infection, or other diseases affecting bile excretion within 3 months prior to screening.
4. Esophageal or gastric variceal bleeding due to portal hypertension within 3 months prior to screening, or history of portosystemic shunt surgery (including Transjugular Intrahepatic Portosystemic Shunt - TIPS) within 6 months prior to screening.
5. History of significant allergy or intolerance to any drug, food, or other substance.
6. History of any clinically significant disease in the neurological, cardiovascular, digestive, respiratory, urinary, endocrine, hematological, immune systems, or any other disease or condition that the investigator believes may affect the trial results.
7. History of surgery that may affect drug absorption, distribution, metabolism, or excretion, or plans for surgery or other reasons requiring hospitalization during the expected study period.
8. Uncontrolled bacterial, viral, parasitic, or fungal infection requiring treatment at the time of screening (except Hepatitis B), or history of severe active infection within 1 month prior to screening.
9. Positive Human Immunodeficiency Virus (HIV) antigen/antibody test at screening. For participants with normal hepatic function: Positive Treponema pallidum antibody. For hepatically impaired participants: Active syphilis.
10. Use of systemic medications with known potential hepatotoxicity for 7 consecutive days or more within 14 days prior to study drug administration.
11. Use of traditional Chinese medicine (herbal medicines, proprietary Chinese medicines), dietary supplements, or vitamins within 14 days prior to study drug administration.
12. Systemic use of moderate or potent CYP3A4 inhibitors (e.g., itraconazole, fluconazole) or moderate or potent CYP3A4 inducers within 14 days prior to study drug administration.
13. Positive urine drug screen or alcohol breath test at screening.
14. Excessive alcohol intake (averaging more than 14 units of alcohol per week) within 3 months prior to screening, or inability to abstain from alcohol during the trial period.
15. Consumption of grapefruit/juice, foods or beverages rich in methylxanthines, engagement in strenuous exercise, or presence of other factors affecting drug absorption, distribution, metabolism, or excretion within 7 days prior to study drug administration, and inability to abstain from these during the hospitalization period.
16. Participation in other investigational drug or medical device clinical trials within 3 months prior to the first dose of the study drug, or participation in 3 or more drug or medical device clinical trials within the past year. If the half-life of the other investigational drug is long, a longer interval is required, at least 5 times the half-life of that drug.
17. Blood donation (or blood loss) ≥ 400 mL, or receipt of blood transfusion or blood products within 3 months prior to screening.
18. History of needle or blood phobia, difficulty with blood collection, or intolerance to venipuncture.
19. Unwillingness or inability to comply with the study procedures outlined in the protocol, or any other reason considered by the investigator as unsuitable for participation in this clinical study.
20. Additional Criteria for Participants with Normal Hepatic Function Only:

1). For participants with normal hepatic function: History of hepatitis, Hepatitis B, or Hepatitis C. History of hepatic impairment, or findings during screening physical examination or laboratory tests suggesting existing or potential hepatic impairment; Positive Hepatitis B Surface Antigen (HBsAg) or positive anti-HCV antibody.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration C(max) | Day 1 to Day 9
  The C(max) of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Time to C(max) [ t(max) ] | Day 1 to Day 9
  The t(max) of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Apparent terminal elimination half-life (t½) | Day 1 to Day 9
  The t½ of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Area under the concentration-time curve from time zero to last time of quantifiable concentration [AUC(last)] | Day 1 to Day 9
  The AUC(last) of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Area under the concentration-time curve from time zero to 192h AUC(0-192h) | Day 1 to Day 9
  The AUC(0-192h) of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Apparent Clearance (CL/F) | Day 1 to Day 9
  The CL/F of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Apparent Volume of distribution (Vz/F) | Day 1 to Day 9
  The Vz/F of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.
Unbound Fraction (fu) | Day 1 to Day 9
  The unbound fraction (fu) of a single dose of olverembatinib in participants with impaired hepatic function and controls with normal hepatic function will be evaluated.

SECONDARY OUTCOMES:
Safety evaluation endpoints | Day1-Day21
  Incidence of treatment-related adverse events, abnormalities in clinical laboratory, vital signs and electrocardiogram (ECG) as assessed by CTCAE v5.0. According to CTCAE v5.0, the number and frequency of adverse events after a single dose of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, M.D.,Ph.D., Principal Investigator — M.D.,Ph.D.; Weifeng Zhao, M.D.,Ph.D., Principal Investigator — The First Affiliated Hospital of Suzhou Medical University
Locations (1):
- The First Affiliated Hospital of Suzhou Medical University, Suzhou, Jiangsu, China